CLINICAL TRIAL: NCT06992570
Title: Identification and Risk Assessment of Mild Traumatic Brain Injury (mTBI) in Czech Armed Forces Soldiers During Specific Training Activities
Brief Title: Risk Assessment of Mild Traumatic Brain Injury in Military Training
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Military University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Michal Soták, Principal Investigator, Charles University, Czech Republic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNIPER-mTBI
Record Dates: First submitted 2025-05-12; First posted 2025-05-28 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Trauma, Brain
Keywords: mTBI; Biomechanics; Military Training
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-Risk Military Training Exposure (Experimental): Active-duty soldiers participating in high-risk training activities, including parachute jumps, high-caliber firearms shooting, artillery blasts, and Close Quarters Battle (CQB) exercises. Participants will undergo real-time biomechanical measurement and biomarker analysis to assess mild traumatic brain injury (mTBI) risk.
  Diagnostic biomarker analysis (GFAP, UCH-L1) Real-time biomechanical monitoring (accelerometers, high-speed cameras)
  Interventions: Diagnostic Test: Quantification of mild trauma brain injury risk; Other: Biomechanical Analysis of Head Impact Forces

INTERVENTIONS:
Diagnostic Test: Quantification of mild trauma brain injury risk — Measure the incidence and severity of mTBI among soldiers engaged in high-risk training activities. (e.g. parachute jumps, high-caliber firearms shooting, artillery fire, explosions). Concentration of brain injury biomarkers (GFAP, UCH-L1) in blood samples collected within 24 hours post-exposure
Other: Biomechanical Analysis of Head Impact Forces — Evaluate the mechanical forces experienced by soldiers during high-risk activities using wearable accelerometers and high-speed video analysis. Peak head acceleration (g-force) and pressure wave analysis during training activities.

SUMMARY:
The SNIPER-TBI study aims to identify and quantify the risk of mild traumatic brain injury (mTBI) in soldiers of the Czech Armed Forces during specific high-risk training activities, including parachute jumps, high-caliber firearms shooting, artillery blasts, and Close Quarters Battle (CQB) exercises. The study will utilize both diagnostic biomarker analysis and experimental biomechanical measurements to assess the physiological impact of these activities on brain health. The ultimate goal is to reduce mTBI incidence, improve operational readiness, and extend the active service duration of soldiers through targeted preventive measures.

DETAILED DESCRIPTION:
The SNIPER-TBI study aims to quantify the risk of mild traumatic brain injury (mTBI) in Czech Armed Forces soldiers during high-risk training activities, including parachute jumps, high-caliber firearms shooting, artillery blasts, and Close Quarters Battle (CQB) exercises. The study combines diagnostic biomarker analysis (GFAP, UCH-L1) and experimental biomechanical measurements using wearable sensors and high-speed cameras. These data will provide critical insights into the forces exerted on the brain during training and help establish exposure limits to minimize long-term neurological impairment. The results will guide the development of protective strategies and enhance soldier readiness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Active-duty military personnel
* Participating in designated high-risk training activities

Exclusion Criteria:

* History of significant brain injury
* Current neurological disorders
* Use of anticoagulant medications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Quantification of mTBI Risk 1 | Up to 24 hours post-exposure
  Measure the severity of mTBI among soldiers engaged in high-risk training activity.
  Concentration of brain injury biomarker glial fibrillary acidic protein (GFAP) in blood sample collected within 24 hours post-exposure. Measured in nanogram per milliliter.
Quantification of mTBI Risk 2 | Up to 24 hours post-exposure
  Measure the severity of mTBI among soldiers engaged in high-risk training activity.
  Concentration of brain injury biomarker ubiquitin carboxyl-terminal hydrolase L1 (UCH-L1) in blood sample collected within 24 hours post-exposure. Measured in nanogram per milliliter.
Biomechanical Analysis of Head Impact Forces 1 | Baseline
  Evaluate the mechanical forces experienced by soldiers during high-risk activity using wearable accelerometers and high-speed video analysis. Peak head acceleration (g-force) will be measured during training activity. Measured in meters per second squared.
Biomechanical Analysis of Head Impact Forces 2 | Baseline
  Evaluate the mechanical forces experienced by soldiers during high-risk activities using wearable accelerometers and high-speed video analysis. Pressure wave during training activity will be analyzed. Measures in Pascal.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Soták, M.D., Ph.D., Principal Investigator — Military University Hospital, Prague
Locations (1):
- Military University Hospital Prague, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to concerns regarding participant confidentiality, data privacy, and the sensitive nature of the study involving military personnel.